CLINICAL TRIAL: NCT05919043
Title: Upper Limb-based Movement Priming for Lower Limb Neuroplasticity & Motor Recovery in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Professor, Physical Therapy, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0070
Record Dates: First submitted 2023-05-01; First posted 2023-06-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Upper limb-based movement priming (UL-priming) (Experimental): The upper limb priming task will include rhythmic, bilateral priming involving the movement of at least one major joint in the upper limbs (shoulder, elbow, wrist).
  Interventions: Other: Upper limb-based movement priming (UL-priming)
- Lower limb-based movement priming (LL-priming) (Active Comparator): Participants will perform rhythmic, symmetric, bilateral plantarflexion and dorsiflexion movements.
  Interventions: Other: Lower limb-based movement priming (LL-priming)
- Sham priming (Sham Comparator): Participants will listen to a 1 Hz metronome for 20 minutes as a form of auditory stimulation during the sham priming session.
  Interventions: Other: Sham priming

INTERVENTIONS:
Other: Upper limb-based movement priming (UL-priming) — Repetitive upper limb movements administered to the beat of a metronome.
  Arms: Upper limb-based movement priming (UL-priming)
Other: Lower limb-based movement priming (LL-priming) — Repetitive lower limb movements administered to the beat of a metronome.
  Arms: Lower limb-based movement priming (LL-priming)
Other: Sham priming — Auditory stimulation.
  Arms: Sham priming

SUMMARY:
The goal of this clinical trial is to to determine the effect of movement-based priming using the upper limbs on lower limb neuroplasticity and behaviors in chronic stroke.

The main questions we aim to answer are:

1. What are the acute effect of UL-priming on lower limb neuroplasticity and motor behaviors in persons with stroke compared to other priming modalities?
2. What are the time effects of UL-priming on neuroplasticity and motor behavior in individuals with stroke?

   In this cross over study, participants will be involved in three priming sessions involving

   - UL-priming using rhythmic, symmetric, bilateral priming involving the movement of at least one major joint in the upper limbs.

   AND

   - Sham priming using auditory stimulation (1 Hz metronome).

   AND

   - Lower-limb movement-based priming using rhythmic, symmetric, dorsiflexion and plantarflexion movements.

   Researchers will compare outcome measures between the different priming sessions.

ELIGIBILITY:
Inclusion Criteria:

* Single, monohemispheric stroke
* Chronic stroke (> 6 months prior)
* Residual hemiparetic gait deficits (e.g., abnormal gait pattern)
* Minimum score of stage 2 on the Chedoke Arm Impairment Scale which includes stage 2, task 3 (facilitated elbow flexion) as one of the stage 2 tasks.

Exclusion Criteria:

* Use of anti-spasticity medications
* Existence of other neurological disorders
* Have brainstem or cerebellar lesions.
* Score of ≥2 on the Modified Ashworth Scale.
* MMSE score of <21, to ensure they will follow instructions.
* Non-English-speaking individuals
* Bone, joint or soft tissue injury
* Uncontrolled medical conditions (such as uncontrolled hypertension, untreated cardiac disease, or untreated pulmonary disease)
* No Motor evoked potentials (MEPs) during TMS

TMS exclusion criteria

* Previous adverse reaction to TMS
* Skull abnormalities or fractures
* Concussion within the prior 6 months
* Unexplained, recurring headaches
* Implanted cardiac pacemaker
* Metal implants in the head or face
* History of seizures or epilepsy
* Use of medications that could alter cortical excitability or increase risk of seizure (e.g., antidepressants, antipsychotics, anxiolytics, anticonvulsants)
* Current pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Corticomotor excitability using transcranial magnetic stimulation (TMS) | Change from baseline to immediately after priming and to 24 hours after priming.
  Single-pulse transcranial magnetic stimulation (TMS) will be used to assess the corticomotor excitability from the tibialis anterior and soleus muscles.
Spinal H-reflex excitability using peripheral nerve stimulation (PNS) | Change from baseline to immediately after priming and to 24 hours after priming.
  Peripheral nerve stimulation (PNS) will be used to assess the H reflexes excitability from the soleus muscles.
Muscle Strength | Change from baseline to immediately after priming and to 24 hours after priming.
  An estimate of maximum ankle muscle force will be obtained for three trials of dorsiflexion and plantarflexion contractions using a force transducer and EMG.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, PT, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Brain Plasticity Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No